CLINICAL TRIAL: NCT06212713
Title: Development and Validation of a Health Behaviour Theory-based Questionnaire to Explore the Willingness of Older Adults and Informal Caregivers to Deprescribe
Brief Title: Developement and Validation of the Health Behavior Questionnaire Towards Deprescribing (HBQtD)
Acronym: HBQtD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Other Study IDs: DEPRESCRIBE
Record Dates: First submitted 2023-10-09; First posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Psychological
Keywords: Older adult; Informal caregiver; Deprescribing; Health behavior theories

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Questionnaire respondents: questionnaire will be administered for validation
  Interventions: Other: Questionnaire administration

INTERVENTIONS:
Other: Questionnaire administration — Questionnaire administration - version older adults and informal caregivers

SUMMARY:
The goal of this observational study is to:

1. develop and validate a health behavior theory-based questionnaire to examine the older adults' and informal caregivers' determinants of deprescribing behavior
2. assess the psychometric properties of this new instrument
3. analyze the moderating influence of health literacy and locus of control on the effect of the determinants on deprescribing intention or behavior.

Participants will be involved in the validating process by completing the questionnaire to be validated, as well as the HLS19_Q12 for health literacy and the MHLC questionnaire for locus of control.

DETAILED DESCRIPTION:
BIBLIOGRAPHIC REFERENCES Prescribing medication is an essential dimension in the care of the older adults (i.e. people aged 60 or 65 and over). However, the ageing process leads to physiological changes that can increase the risk of adverse drug events, and inappropriate polypharmacy can contribute to drug-drug interactions, lower medication adherence, significant costs to both the patient and the healthcare system, and also reduce people's ability to perform activities of daily living.

Therefore, it is important thinking about deprescription, defined by Reeve et al. (2022) as "a planned/ supervised process of dose reduction or the stopping of medicines that may be causing harm or conferring no additional benefit".

As implementation deprescribing requires a complexes changes to established patters of behaviors, understanding the cognitive mechanisms underlying patient's and caregiver's behavior with respect to deprescribing, seems essential to improve the collaborative work between the patient, or even the caregivers, and the health professionals, to achieve the best health outcomes for the patient.

In reality, health behavior theories provides a series of concepts deriving from social, cognitive and motivational psychology, that can be useful in understanding why people behave in certain ways in relation to their health.

Screening Tools The patients' attitudes towards deprescribing (PATD) questionnaire, and its revised version questionnaire (rPATD), and Beliefs about Medicines Questionnaire (specific section) (BMQ-Specific) are 2 instruments widely used. However, this questionnaires don't consider critical domains that can be relevant to deprescribing, such as self-efficacy beliefs, outcome expectations, subjective norms, health goals, environmental barriers and enablers, among others.

Hypothesis The investigators hypothesise that some of the gaps in existing tools will be filled by using health behaviour concepts in the development of an assessment tool.

STUDY DESIGN AND METHODOLOGY APPLIED Type of study: Questionnaire development and validation - older adult and informal caregiver version

Study configuration The initial questionnaire was developed considering the results of a previous systematic review (article currently being written), which was intended to identify (concepts included in) behavioral health theories (HBTs) that explain older adults' and informal caregivers' deprescribing intention and/or their actual deprescribing behavior, as well as the rPATD questionnaire and BMQ questionnaire.

The initial version for informal caregivers was developed by modifying the wording of the items, in the version for the older adults, adapting them for informal caregivers.

Another two questionnaires will be used in this study: one that measure health literacy (HLS19_Q12) and another one that assess the locus of control (Multidimensional Health Locus of control scale, MHLC).

The development and validation of the questionnaire comprise 4 main steps:

1. Item Development
2. Preliminary pilot testing

   1. Colleagues questionnaire feedback
   2. "Cognitive pre-test" performed with older adults and informal caregivers to check the linguistic and analytical construction of the items,
   3. First round with healthcare professionals and second round with older adults and informal carers for a self-administered questionnaire and focus group.
3. Pre-test of the questionnaire - older adult and informal caregiver version
4. Validation of the questionnaire - older adult and informal carer versions, using exploratory factor analysis

Strategies for recruiting participants To recruit participants, several organisations and institutions will be contacted.

Data Management Responsibilities The two questionnaire versions will be either a paper version for self-administration and an electronic version available online.

DISSEMINATION OF RESULTS AND PUBLICATION POLICY The progress and results of this study will be discussed with the Di-Prescribe research team. At the end of the study, a scientific publication will be written by the co-investigator (Sara Alves Jorge) under the supervision of the sponsor representative and Prof Van den Broucke. A paper will also be written for publication in a peer-journal. Acknowledgements will be made to all those who will make this work possible, including healthcare professionals, the different institutions and organizations that will be contacted, as well as the older adults and informal caregivers who will take part in the study. In addition, some people who will be indirectly involved, in particular by giving support and guidance, will also be recognized.

ELIGIBILITY:
Inclusion Criteria:

Older adults

* Age 60 years or older;
* Taking at least 5 medications daily;
* Having at least one chronic condition.

Informal caregivers

* They self-identified as a caregiver (defined as having any role in a family member or friend's management of health and/ or medication management) of an older adult who has 60 years old or older, that are taking at least 5 medications daily;
* The care recipient lived in the community (at home with or without the caregiver) or in a NH.

Exclusion Criteria:

Older adults

* Suffering from psychiatric trouble;
* Past or present drug or alcohol dependency;
* Having a terminal illness;
* Inability to complete a written questionnaire in French due to a functional or cognitive impairment;
* Inability to understand and express oneself in French.

Informal cariegivers

* Caregiver age under 18 years old;
* Caregivers who are paid for the care they provide;
* Caregiver inability to give consent and complete a written questionnaire in French;
* Caregiver inability to understand and speak in French.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: For the purposes of this study, older adult are people aged 60 or older. Take at least 5 regular medications: the ageing process is often accompanied by an increasing burden of chronic illness, and consequently by chronic medication use that can lead to polypharmacy, defined as taking 5 or more medications.
  In this study informal caregiver refers to a family member, a friend that provide care or support to a dependent older person with physical or cognitive functions declines. The relationship between the informal caregiver and the care recipient is based on solidarity. Therefore, in this study those who provided informal care are: (a) working-age adults who care for older parents with disabilities, family members, neighbors or friends; (b) people of retirement age or older who care for their partner, family members, neighbors or friends
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Validity and reliability of the measurement tool - HBQtD | Throughout the entire study, approximately during 9 months
  Questionnaire administration (HBQtD) for psychometric analyse
Correlation between deprescribing intention and behavior and deprescribing determinants using HBQtD questionnaire | Throughout the entire study, approximately during 9 months
  Questionnaire administration (HBQtD) and regression analysis will be performed

SECONDARY OUTCOMES:
Moderating effect of health literacy using HLS19_Q12 | Throughout the entire study, approximately during 9 months
  HLS19_Q12 questionnaire administration and regression analysis will be performed
Moderating effect of locus of control using Multidimensional Health locus of control scale (MHLC) | Throughout the entire study, approximately during 9 months
  MHLC scale administration and regression analysis will be performed

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Van den Broucke, PhD, Principal Investigator — Université Catholique de Louvain
Locations (1):
- UCLouvain, Louvain-la-Neuve, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abouzaid, S., Willemse, E., Remmen, R., Schmitz, O., Macq, J., Declercq, A., Arnaut, C., Forest, M., Denis, A., Vinck, I., Defourny, N., & Farfan-Portet, M. (s. d.). SUPPORT FOR INFORMAL CAREGIVERS - AN EXPLORATORY ANALYSIS.
- [Background] Aithal, A., & Aithal, P. S. (2020). Development and Validation of Survey Questionnaire & Experimental Data - A Systematical Review-based Statistical Approach (SSRN Scholarly Paper No 3724105). https://doi.org/10.2139/ssrn.3724105
- [Background] Ajzen, I. (1991). The Theory of Planned Behavior.
- [Background] Ajzen, I., & Madden, T. J. (1986). Prediction of goal-directed behavior : Attitudes, intentions, and perceived behavioral control. Journal of Experimental Social Psychology, 22(5), 453-474. https://doi.org/10.1016/0022-1031(86)90045-4
- [Background] Bandura A. Health promotion by social cognitive means. Health Educ Behav. 2004 Apr;31(2):143-64. doi: 10.1177/1090198104263660. PMID 15090118
- [Background] Baumgartner AD, Clark CM, LaValley SA, Monte SV, Wahler RG Jr, Singh R. Interventions to deprescribe potentially inappropriate medications in the elderly: Lost in translation? J Clin Pharm Ther. 2020 Jun;45(3):453-461. doi: 10.1111/jcpt.13103. Epub 2019 Dec 24. PMID 31873955
- [Background] Beers MH. Explicit criteria for determining potentially inappropriate medication use by the elderly. An update. Arch Intern Med. 1997 Jul 28;157(14):1531-6. PMID 9236554
- [Background] Chock YL, Wee YL, Gan SL, Teoh KW, Ng KY, Lee SWH. How Willing Are Patients or Their Caregivers to Deprescribe: a Systematic Review and Meta-analysis. J Gen Intern Med. 2021 Dec;36(12):3830-3840. doi: 10.1007/s11606-021-06965-5. Epub 2021 Jun 25. PMID 34173200
- [Background] Clark LA, Watson D. Constructing validity: New developments in creating objective measuring instruments. Psychol Assess. 2019 Dec;31(12):1412-1427. doi: 10.1037/pas0000626. Epub 2019 Mar 21. PMID 30896212
- [Background] Doval E, Viladrich C, Angulo-Brunet A. Coefficient Alpha: The Resistance of a Classic. Psicothema. 2023 Feb;35(1):5-20. doi: 10.7334/psicothema2022.321. PMID 36695846
- [Background] Dunn TJ, Baguley T, Brunsden V. From alpha to omega: a practical solution to the pervasive problem of internal consistency estimation. Br J Psychol. 2014 Aug;105(3):399-412. doi: 10.1111/bjop.12046. Epub 2013 Aug 6. PMID 24844115
- [Background] Elsesser, K., & Sartory, G. (1998). OUTCOME PREDICTORS OF BENZODIAZEPINE WITHDRAWAL. Behavioural and Cognitive Psychotherapy, 26(3), 209-217. https://doi.org/10.1017/S135246589800023X
- [Background] Gabauer J. CE: Mitigating the Dangers of Polypharmacy in Community-Dwelling Older Adults. Am J Nurs. 2020 Feb;120(2):36-42. doi: 10.1097/01.NAJ.0000654312.14385.3d. PMID 31977416
- [Background] Gehlert, S., & Ward, T. S. (2019). Theories of Health Behavior. In S. Gehlert & T. Browne (Éds.), Handbook of Health Social Work (1re éd., p. 143-163). Wiley. https://doi.org/10.1002/9781119420743.ch7
- [Background] Gillespie R, Mullan J, Harrison L. Managing medications: the role of informal caregivers of older adults and people living with dementia. A review of the literature. J Clin Nurs. 2014 Dec;23(23-24):3296-308. doi: 10.1111/jocn.12519. Epub 2013 Dec 20. PMID 24354583
- [Background] Gillespie R, Mullan J, Harrison L. Attitudes towards deprescribing and the influence of health literacy among older Australians. Prim Health Care Res Dev. 2019 Jun 20;20:e78. doi: 10.1017/S1463423618000919. PMID 32799987
- [Background] Godin, G. (1991). L'éducation pour la santé : Les fondements psycho-sociaux de la définition des messages éducatifs. Sciences Sociales et Santé, 9(1), 67-94. https://doi.org/10.3406/sosan.1991.1185
- [Background] Hanlon JT, Schmader KE. The Medication Appropriateness Index: A Clinimetric Measure. Psychother Psychosom. 2022;91(2):78-83. doi: 10.1159/000521699. Epub 2022 Feb 14. No abstract available. PMID 35158365
- [Background] Harris PA, Taylor R, Minor BL, Elliott V, Fernandez M, O'Neal L, McLeod L, Delacqua G, Delacqua F, Kirby J, Duda SN; REDCap Consortium. The REDCap consortium: Building an international community of software platform partners. J Biomed Inform. 2019 Jul;95:103208. doi: 10.1016/j.jbi.2019.103208. Epub 2019 May 9. PMID 31078660
- [Background] Hinkin, T. R. (1998). A Brief Tutorial on the Development of Measures for Use in Survey Questionnaires. Organizational Research Methods, 1(1), 104-121. https://doi.org/10.1177/109442819800100106
- [Background] Horne, R., Weinman, J., & Hankins, M. (1999). The Beliefs About Medicines Questionnaire : The Development and Evaluation of a New Method for Assessing the Cognitive Representation of Medication. Psychology & Health, 14(1), 1. https://doi.org/10.1080/08870449908407311
- [Background] Koo TK, Li MY. A Guideline of Selecting and Reporting Intraclass Correlation Coefficients for Reliability Research. J Chiropr Med. 2016 Jun;15(2):155-63. doi: 10.1016/j.jcm.2016.02.012. Epub 2016 Mar 31. PMID 27330520
- [Background] Lachman ME. Locus of control in aging research: a case for multidimensional and domain-specific assessment. Psychol Aging. 1986 Mar;1(1):34-40. doi: 10.1037//0882-7974.1.1.34. PMID 3267376
- [Background] Landis JR, Koch GG. The measurement of observer agreement for categorical data. Biometrics. 1977 Mar;33(1):159-74. PMID 843571
- [Background] Linsky A, Simon SR, Bokhour B. Patient perceptions of proactive medication discontinuation. Patient Educ Couns. 2015 Feb;98(2):220-5. doi: 10.1016/j.pec.2014.11.010. Epub 2014 Nov 20. PMID 25435516
- [Background] Martin P, Tamblyn R, Ahmed S, Tannenbaum C. A drug education tool developed for older adults changes knowledge, beliefs and risk perceptions about inappropriate benzodiazepine prescriptions in the elderly. Patient Educ Couns. 2013 Jul;92(1):81-7. doi: 10.1016/j.pec.2013.02.016. Epub 2013 Mar 29. PMID 23541509
- [Background] McCoach, D. B., Gable, R. K., & Madura, J. P. (2013). Instrument Development in the Affective Domain : School and Corporate Applications. Springer. https://doi.org/10.1007/978-1-4614-7135-6
- [Background] McDonald, R. P. (1999). Test Theory : A Unified Treatment. Psychology Press. https://doi.org/10.4324/9781410601087
- [Background] Muhlack DC, Hoppe LK, Weberpals J, Brenner H, Schottker B. The Association of Potentially Inappropriate Medication at Older Age With Cardiovascular Events and Overall Mortality: A Systematic Review and Meta-Analysis of Cohort Studies. J Am Med Dir Assoc. 2017 Mar 1;18(3):211-220. doi: 10.1016/j.jamda.2016.11.025. Epub 2017 Jan 26. PMID 28131719
- [Background] Olsson IN, Runnamo R, Engfeldt P. Medication quality and quality of life in the elderly, a cohort study. Health Qual Life Outcomes. 2011 Nov 3;9:95. doi: 10.1186/1477-7525-9-95. PMID 22054205
- [Background] O'Donnell LK, Ibrahim K. Polypharmacy and deprescribing: challenging the old and embracing the new. BMC Geriatr. 2022 Sep 7;22(1):734. doi: 10.1186/s12877-022-03408-6. No abstract available. PMID 36068485
- [Background] Oktora MP, Edwina AE, Denig P. Differences in Older Patients' Attitudes Toward Deprescribing at Contextual and Individual Level. Front Public Health. 2022 Feb 11;10:795043. doi: 10.3389/fpubh.2022.795043. eCollection 2022. PMID 35223732
- [Background] Page AT, Clifford RM, Potter K, Schwartz D, Etherton-Beer CD. The feasibility and effect of deprescribing in older adults on mortality and health: a systematic review and meta-analysis. Br J Clin Pharmacol. 2016 Sep;82(3):583-623. doi: 10.1111/bcp.12975. Epub 2016 Jun 13. PMID 27077231
- [Background] Parekh N, Ali K, Davies K, Rajkumar C. Can supporting health literacy reduce medication-related harm in older adults? Ther Adv Drug Saf. 2018 Mar;9(3):167-170. doi: 10.1177/2042098618754482. Epub 2018 Feb 9. No abstract available. PMID 29492245
- [Background] Parker G, Shahid N, Rappon T, Kastner M, Born K, Berta W. Using theories and frameworks to understand how to reduce low-value healthcare: a scoping review. Implement Sci. 2022 Jan 20;17(1):6. doi: 10.1186/s13012-021-01177-1. PMID 35057832
- [Background] Pazan F, Wehling M. Polypharmacy in older adults: a narrative review of definitions, epidemiology and consequences. Eur Geriatr Med. 2021 Jun;12(3):443-452. doi: 10.1007/s41999-021-00479-3. Epub 2021 Mar 10. PMID 33694123
- [Background] Pelikan JM, Link T, Strassmayr C, Waldherr K, Alfers T, Boggild H, Griebler R, Lopatina M, Miksova D, Nielsen MG, Peer S, Vrdelja M; HLS19 Consortium of the WHO Action Network M-POHL. Measuring Comprehensive, General Health Literacy in the General Adult Population: The Development and Validation of the HLS19-Q12 Instrument in Seventeen Countries. Int J Environ Res Public Health. 2022 Oct 29;19(21):14129. doi: 10.3390/ijerph192114129. PMID 36361025
- [Background] Petein C, Spinewine A, Laroche ML, Niquille A, Henrard S. Adaptation and validation of the revised Patients' Attitudes towards Deprescribing (rPATD) questionnaire for benzodiazepine receptor agonists. Res Social Adm Pharm. 2023 Sep;19(9):1278-1285. doi: 10.1016/j.sapharm.2023.05.010. Epub 2023 Jun 8. PMID 37301641
- [Background] Prochaska JO, DiClemente CC. Stages and processes of self-change of smoking: toward an integrative model of change. J Consult Clin Psychol. 1983 Jun;51(3):390-5. doi: 10.1037//0022-006x.51.3.390. No abstract available. PMID 6863699
- [Background] Prochaska JO, Velicer WF. The transtheoretical model of health behavior change. Am J Health Promot. 1997 Sep-Oct;12(1):38-48. doi: 10.4278/0890-1171-12.1.38. PMID 10170434
- [Background] Reeve E, Low LF, Shakib S, Hilmer SN. Development and Validation of the Revised Patients' Attitudes Towards Deprescribing (rPATD) Questionnaire: Versions for Older Adults and Caregivers. Drugs Aging. 2016 Dec;33(12):913-928. doi: 10.1007/s40266-016-0410-1. PMID 27785734
- [Background] Reeve E, Shakib S, Hendrix I, Roberts MS, Wiese MD. Development and validation of the patients' attitudes towards deprescribing (PATD) questionnaire. Int J Clin Pharm. 2013 Feb;35(1):51-6. doi: 10.1007/s11096-012-9704-5. Epub 2012 Oct 9. PMID 23054137
- [Background] Reeve E, To J, Hendrix I, Shakib S, Roberts MS, Wiese MD. Patient barriers to and enablers of deprescribing: a systematic review. Drugs Aging. 2013 Oct;30(10):793-807. doi: 10.1007/s40266-013-0106-8. PMID 23912674
- [Background] Reeve E, Wolff JL, Skehan M, Bayliss EA, Hilmer SN, Boyd CM. Assessment of Attitudes Toward Deprescribing in Older Medicare Beneficiaries in the United States. JAMA Intern Med. 2018 Dec 1;178(12):1673-1680. doi: 10.1001/jamainternmed.2018.4720. PMID 30326004
- [Background] Reeve J, Maden M, Hill R, Turk A, Mahtani K, Wong G, Lasserson D, Krska J, Mangin D, Byng R, Wallace E, Ranson E. Deprescribing medicines in older people living with multimorbidity and polypharmacy: the TAILOR evidence synthesis. Health Technol Assess. 2022 Jul;26(32):1-148. doi: 10.3310/AAFO2475. PMID 35894932
- [Background] Rogers RW. A Protection Motivation Theory of Fear Appeals and Attitude Change1. J Psychol. 1975 Sep;91(1):93-114. doi: 10.1080/00223980.1975.9915803. PMID 28136248
- [Background] Roux B, Rakheja B, Sirois C, Niquille A, Petein C, Ouellet N, Spinewine A, Sibille FX, Laroche ML. Attitudes and beliefs of older adults and caregivers towards deprescribing in French-speaking countries: a multicenter cross-sectional study. Eur J Clin Pharmacol. 2022 Oct;78(10):1633-1646. doi: 10.1007/s00228-022-03368-1. Epub 2022 Jul 27. PMID 35896803
- [Background] Scott S, Wright DJ, Bhattacharya D. The role of behavioural science in changing deprescribing practice. Br J Clin Pharmacol. 2021 Jan;87(1):39-41. doi: 10.1111/bcp.14595. Epub 2020 Nov 5. No abstract available. PMID 33037662
- [Background] Seewoodharry M, Khunti K, Davies MJ, Gillies C, Seidu S. Attitudes of older adults and their carers towards de-prescribing: A systematic review. Diabet Med. 2022 Jul;39(7):e14801. doi: 10.1111/dme.14801. Epub 2022 Feb 15. PMID 35118700
- [Background] Spinewine A, Schmader KE, Barber N, Hughes C, Lapane KL, Swine C, Hanlon JT. Appropriate prescribing in elderly people: how well can it be measured and optimised? Lancet. 2007 Jul 14;370(9582):173-184. doi: 10.1016/S0140-6736(07)61091-5. PMID 17630041
- [Background] Steinman MA. Polypharmacy-Time to Get Beyond Numbers. JAMA Intern Med. 2016 Apr;176(4):482-3. doi: 10.1001/jamainternmed.2015.8597. No abstract available. PMID 26999383
- [Background] Strauss ME, Smith GT. Construct validity: advances in theory and methodology. Annu Rev Clin Psychol. 2009;5:1-25. doi: 10.1146/annurev.clinpsy.032408.153639. PMID 19086835
- [Background] Trizano-Hermosilla I, Alvarado JM. Best Alternatives to Cronbach's Alpha Reliability in Realistic Conditions: Congeneric and Asymmetrical Measurements. Front Psychol. 2016 May 26;7:769. doi: 10.3389/fpsyg.2016.00769. eCollection 2016. PMID 27303333
- [Background] Tsang S, Royse CF, Terkawi AS. Guidelines for developing, translating, and validating a questionnaire in perioperative and pain medicine. Saudi J Anaesth. 2017 May;11(Suppl 1):S80-S89. doi: 10.4103/sja.SJA_203_17. PMID 28616007
- [Background] Turner JP, Martin P, Zhang YZ, Tannenbaum C. Patients beliefs and attitudes towards deprescribing: Can deprescribing success be predicted? Res Social Adm Pharm. 2020 Apr;16(4):599-604. doi: 10.1016/j.sapharm.2019.07.007. Epub 2019 Jul 10. PMID 31303479
- [Background] Wallston KA, Wallston BS, DeVellis R. Development of the Multidimensional Health Locus of Control (MHLC) Scales. Health Educ Monogr. 1978 Spring;6(2):160-70. doi: 10.1177/109019817800600107. PMID 689890
- [Background] Weir KR, Ailabouni NJ, Schneider CR, Hilmer SN, Reeve E. Consumer Attitudes Towards Deprescribing: A Systematic Review and Meta-Analysis. J Gerontol A Biol Sci Med Sci. 2022 May 5;77(5):1020-1034. doi: 10.1093/gerona/glab222. PMID 34390339
- [Background] Wolff JL, Boyd CM. A Look at Person- and Family-Centered Care Among Older Adults: Results from a National Survey [corrected]. J Gen Intern Med. 2015 Oct;30(10):1497-504. doi: 10.1007/s11606-015-3359-6. Epub 2015 May 2. PMID 25933625
- [Background] Yong, A. G., & Pearce, S. (2013). A Beginner's Guide to Factor Analysis : Focusing on Exploratory Factor Analysis.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-11): https://cdn.clinicaltrials.gov/large-docs/13/NCT06212713/Prot_SAP_000.pdf
  • Informed Consent Form (2023-08-14): https://cdn.clinicaltrials.gov/large-docs/13/NCT06212713/ICF_001.pdf